CLINICAL TRIAL: NCT01761344
Title: Intraoperative Analysis of Cortisol During Adrenal Vein Catheterization and Sampling in Patients With Primary Hyperaldosteronism.
Brief Title: Intraoperative Analysis of Cortisol During Adrenal Vein Sampling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012/1856
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Primary Hyperaldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraoperative measurement of cortisol (Experimental): Intervention: During a routine procedure intraoperative cortisol is measured. Upon unsuccessful sampling, the sampling will be repeated.
  Interventions: Other: Intraoperative cortisol measurement.

INTERVENTIONS:
Other: Intraoperative cortisol measurement. — Levels of cortisol in blood samples will be determined using a rapid cortisol assay. This is not standard procedure

SUMMARY:
Aldosterone is a hormone produced in the adrenals that helps regulate the salt balance and blood pressure. Primary hyperaldosteronism is one of the main endocrine causes of secondary hypertension. The overproduction of aldosteron might in some cases be due to unilateral hyperplasia of the adrenal cortex or a unilateral aldosterone-producing adenoma. In these cases the adrenal can be removed and the patient cured of hypertension. The clinical evaluation of patients with confirmed primary hyperaldosteronism therefore includes selective sampling of blood from the adrenal veins to determine lateralization of overproduction. This is executed as an interventional radiological procedure.

The adrenal vein sampling is challenging, and success is determined by measuring another adrenal hormone named cortisol in the blood samples as a marker of a correctly drawn sample. By routine laboratory assays the procedure is evaluated after the patient has been discharged from the hospital. In the study a rapid assay of cortisol will be evaluated, allowing the radiologist to draw new samples during the same procedure if the first set of samples is unsuccessful. The study hypothesis is that intraoperative measurement of cortisol is a useful tool to evaluate successful sampling, and that fewer patients will need a repeated procedure.

ELIGIBILITY:
Inclusion Criteria:

* Primary hyperaldosteronism
* Motivated for surgery if applicable
* Able to give informed consent

Exclusion Criteria:

* Not able to give informed consent
* Severe kidney failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Representative blood sample from adrenal veins bilaterally. | Intraoperatively
  Patients where the drawn blood from both adrenal veins is representative is the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Mellgren, MD.PhD, Study Chair — Hormonlaboratoriet, Haukeland Universitetssykehus
Locations (1):
- Haukeland University Hospital, Bergen, Hordaland, Norway